CLINICAL TRIAL: NCT05206968
Title: Scoring System of Structural Damage for the Hip in Juvenile Idiopathic Arthritis
Acronym: hip index
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, lassoued ferjani Hanene, Assistant professor, University Tunis El Manar
Other Study IDs: 5981
Record Dates: First submitted 2022-01-12; First posted 2022-01-25 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Juvenile Idiopathic Arthritis Hip

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: pelvic radiograph — Patients with hip involvement underwent a pelvic radiograph

SUMMARY:
Juvenile idiopathic arthritis (JIA) is a chronic inflammatory disease in children affecting mobility and physical function. The hip involvement represents a frequent complication in JIA patients. The assessment of hip damage becomes a mandatory step in disease monitoring. However, radiological scoring was not standardized. This study aimed to compare the two scoring systems previously proposed, examine their repeatability and their intra and inter agreement.

ELIGIBILITY:
Inclusion Criteria:

* All included patient followed the ILAR criteria of JIA and have a hip involvement. This later was defined as the presence of rang motion limitation, and abnormal findings in pelvic radiographic, or ultrasound or MRI in the coxo-femoral joint.

Exclusion Criteria:

* The presence of a contraindication to the performance of conventional radiography any disease affecting cognition Patients who have had surgery on the hip

Ages: 4 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: General data demographics , disease characteristics [symptom duration, disease presentation, JIA subtypes, Antigen(HLA) B27 positivity)], disease activity: Juvenile arthritis disease activity (JADAS), were collected.
  All patients underwent a posteroanterior pelvic radiograph
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
intermodality agreement | 6 months
  mesuring the intermodality agreement between two scoring system: the The Childhood Arthritis Radiographic Score of the Hip (CARSH) and the new radiographic scoring system for growth abnormalities and structural change in children with juvenile idiopathic arthritis of the hip

SECONDARY OUTCOMES:
interreader agreement | 3 months
  mesuring the interreader agreement between two experimented pediatric rheumatologist for the assessement of structurla damage in JIA hip

CONTACTS AND LOCATIONS:
Locations (1):
- Kassab institute of orthopedics, Manouba, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Maatallah K, Lassoued Ferjani H, Ben Nessib D, Dghaies A, Kharrat L, Majdoub F, Kaffel D, Hamdi W. Can pediatric rheumatologists apply available hip scoring systems in daily practice for juvenile idiopathic arthritis? Front Pediatr. 2025 Mar 28;13:1436200. doi: 10.3389/fped.2025.1436200. eCollection 2025. PMID 40224384